CLINICAL TRIAL: NCT06395597
Title: Variability of Healthy People and People After Stroke Results in the Nine Hole Peg Test
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Rybářová, Occupational therapist, Charles University, Czech Republic
Other Study IDs: 23/4
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Motor Activity
Keywords: Nine Hole Peg Test; stroke; Czech Extended Version of Manual for the Nine Hole Peg Test
MeSH Terms: conditions — Motor Activity; Stroke | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- People after stroke: Czech people after stroke, aged 20 - 64 years
  Interventions: Diagnostic Test: Nine Hole Peg Test
- Healthy population: Czech healthy people, aged 20 - 64 years
  Interventions: Diagnostic Test: Nine Hole Peg Test

INTERVENTIONS:
Diagnostic Test: Nine Hole Peg Test — 3 attempts of each subtest of the Nine Hole Peg Test performed according to the Czech Extended Version of Manual for the Nine Hole Peg Test; questionnaire
  Other Names: questionnaire

SUMMARY:
Main aim of the study is to find out how many attempts of each subtest in the Nine Hole Peg Test should be done in clinical practice during testing people after stroke who are 20-64 years old.

ELIGIBILITY:
Inclusion Criteria:

* age: 20-64 years (inclusive)
* hospitalized patient in Rehabilitation Centre Kladruby
* women and men with Czech as their mother tongue
* signed Informed consent
* ability to maintain a stable sitting position for the duration necessary for testing
* comprehension of verbal instructions and recordings for the Nine Hole Peg Test

Exclusion Criteria:

* inability to successfully complete a pilot attempt of the Nine Hole Peg Test using the right and left hand
* severe spastic paresis of the upper limb, which would make the test impossible
* plegia of the upper limb
* failure to complete the test to visual or hearing impairment
* inability to understand verbal instructions
* inability to maintain attention during testing
* severe attention deficit disorder
* neglect syndrome
* fatigue
* external factors that prevent the complete completion of the test

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Czech healthy people and Czech people after stroke
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
results from the Nine Hole Peg Test | 30 minutes
  time

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Rybářová, Mgr., Principal Investigator — Charles University, Czech Republic
Locations (2):
- Czechia (2):
  - Rehabilitační ústav Kladruby, Kladruby
  - Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: No